CLINICAL TRIAL: NCT00974285
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trials on the Effect of Immunity 1 (Fuzheng 1) on Immune Reconstitution of HIV Patients
Brief Title: Clinical Trials on the Effect of Immunity 1 (Fuzheng 1) on Immune Reconstitution of HIV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: WANG, Jie/Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.07.16-3
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-09

CONDITIONS: Acquired Immune Deficiency Syndrome Virus; HIV Infections
Keywords: AIDS; complementary therapies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fuzheng 1 (Active Comparator): Immunity 1 (Fuzheng 1), 8.75g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Fuzheng 1
- Placebo (Placebo Comparator): Placebo, 8.75g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fuzheng 1 — Immunity 1 (Fuzheng 1), 8.75g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Fuzheng 1
Drug: Placebo — Placebo, 8.75g twice a day, half an hour before breakfast and dinner, mixing with water, for six successive cycles of 30 days.
  Arms: Placebo

SUMMARY:
The average period of asymptomatic HIV-infection is 8 years, at this stage, CD4+ T lymphocyte count was reduced gradually at the rate of 50~100cells/ul/year. When the CD4 T lymphocyte count dropped below 350cells/ul and viral load increased to 105 in AIDS patients, HAART will be carried out. But, CD4 T lymphocyte was 350~550 cells/ul, there is no intervention measures.

DETAILED DESCRIPTION:
* The average period of asymptomatic HIV-infection is 8 years, at this stage, CD4+ T lymphocyte count was reduced gradually at the rate of 50~100cells/ul/year. When the CD4 T lymphocyte count dropped below 350cells/ul and viral load increased to 105 in AIDS patients, HAART will be carried out. But, CD4 T lymphocyte was 350~550 cells/ul, there is no intervention measures.
* Immunity 1 (Fuzheng 1) is composed of herbs which have tonic and detoxific function. The long-term clinical application has proved the safety and effect. It can improve the symptoms and signs in AIDS patients with the effective rate of 70% and can significantly improve the quality of life. It can also improve and stabilize immune function and inhibit viral replication. The basis study have shown that Immunity 1 (Fuzheng 1) can inhibit viral replication from multi-target, multi-link, enhance immune function, increase the secretion of IL-2, IFN-γ, participate in immune regulation effect, enhance NK cell activity, promote CD3+CD4+T cell proliferation and increase macrophage phagocytes capacity.
* Through the clinical trials, we are going to evaluate the efficacy and safety of Immunity 1 (Fuzheng 1) on immune reconstitution of HIV patients in WHOⅠ、II period.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody-positive, confirmed by Western Blot test
* CD 4 counts> 350 cells / ul and <550 cells / ul
* Age ≥ 18 years old and ≤ 70 years old
* Voluntary participated in this study, signed informed consent form, and could be followed-up

Exclusion Criteria:

* Patients in WHO clinical stage Ⅲ, Ⅳ
* Participated in clinical trials of other drugs within one month before the experiment
* Received antiretroviral therapy or are anti-HIV drugs such as nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs) and fusion-inhibiting agent (FIs), integrase inhibitors, inhibitors penetration within one month before the experiment
* Received immunomodulatory treatment within one month before the experiment Liver and kidney dysfunction (AST, ALT, T-BIL ≥2 times of upper limit of the reference value or creatinine ≥ 2 times of the upper limit of reference value)
* Patients with obvious active diseases in respiratory system, digestive system, circulatory system, blood system, neuroendocrine system, or genitourinary system diseases
* Persons suffering from autoimmune diseases
* Cancer patients which need chemotherapy
* Pregnant or lactating women, and did not use safe contraceptive measures for women of child-bearing age, as well as the male that can not take a reasonable method of contraception in trial period
* Hypersensitive people
* Patients with dysgnosia or language barriers, which can not fully understand the test or cooperate well

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood CD3+ CD4+ counts | 6 months

SECONDARY OUTCOMES:
Immune reconstitution efficiency | 6 months
Viral load | 6 months
Clinical symptoms and signs | 6 months
KPS score | 6 months
Quality of life score | 6 months
Safety evaluation | 6 months
Economic evaluation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie WANG, MD, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Jie, WANG, Beijing, Beijing Municipality, China